CLINICAL TRIAL: NCT01113385
Title: Effect of Oral Galactose on the Level of Focal Sclerosis Permeability Factor and Proteinuria in Children With Steroid Resistant Nephrotic Syndrome: A Pilot Study
Brief Title: Oral Galactose in Children With Steroid Resistant Nephrotic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: National Kidney Foundation, United States (Other)
Responsible Party: Principal Investigator, Asha Moudgil, Professor of Pediatrics, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4657
Record Dates: First submitted 2010-04-28; First posted 2010-04-29 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Focal Segmental Glomerulosclerosis; Steroid Resistant Nephrotic Syndrome
Keywords: Nephrotic syndrome; Focal Segmental glomerulosclerosis; FSGS; Minimal change; Steroid resistant; Pediatric; Proteinuria; Galactose; FSPF
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Nephrotic Syndrome; Proteinuria | interventions — Galactose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Galactose (Experimental): Oral galactose will be given at a dose of 0.2gm/kg/dose twice a day (BID) to a maximum of 15 gm BID for a period of 16 weeks.
  Interventions: Drug: D-Galactose

INTERVENTIONS:
Drug: D-Galactose — Oral galactose will be initiated at a dose of 0.2gm/kg/dose twice daily to a maximum of 15 gm BID for a period of 4 months. The prescribed dose of D-galactose powder will be dispensed to subjects in packets, mixed with 4 ounces of water, and consumed orally.
  Other Names: Galactose

SUMMARY:
Focal Segmental Glomerulosclerosis (FSGS) is a devastating kidney disease which is difficult to treat and carries a poor prognosis, with 50% of affected children progressing to end stage renal disease (ESRD). The purpose of this study is to investigate oral galactose as a benign treatment for FSGS in children. The investigators hypothesize that galactose, a simple milk sugar thought to bind to the protein factor (FSPF) that causes FSGS thereby inactivating it and stopping it from damaging the kidney, resulting in a reduction in glomerular permeability to albumin and decrease in proteinuria in children with nephrotic syndrome secondary to FSGS.

DETAILED DESCRIPTION:
RESEARCH PLAN

A: Primary aims:

1. Determine the effect of 4 months of oral galactose administration on the level of FSPF in children with steroid resistant FSGS
2. Determine the effect of 4 months of oral galactose administration on the first morning urine protein to creatinine (urine protein: creatinine) ratio and serum albumin level in children with steroid resistant FSGS.

B: Secondary aims:

1. Determine the effect of 4 months of oral galactose administration on dose of immunosuppressive medication.
2. Assess first morning urine protein: creatinine ratio, serum albumin level, and change in immunosuppression dose at 3 months after discontinuation of oral galactose therapy.

B.Background and Significance

Idiopathic nephrotic syndrome (NS) in children is most commonly due to minimal change nephrotic syndrome and can be successfully treated with steroid therapy. However 10-15% of children with nephrotic syndrome are diagnosed with FSGS, which is resistant to steroid therapy and many other immunosuppressive drugs, and is associated with poor outcome. Approximately 50% of patients with FSGS progress to ESRD within 5-10 years and in about 30% of children, FSGS can recur after transplantation.(1) African-American children are at significantly higher risk for FSGS.(2) Recent studies indicate that primary FSGS is a heterogeneous disorder caused by genetic mutations in nearly a third of cases and as yet undefined immunological defects in the remaining cases.(3) Immune mediated FSGS has been associated with a circulating permeability factor, which is thought to increase glomerular permeability to albumin, leading to proteinuria and contributes to sclerotic lesions in FSGS. Presence of the FSPF is defined as permeability activity >0.5. (4) Current therapies for FSGS include plasmapheresis and many immunosuppressive agents that include cyclosporine, tacrolimus, mycophenolate mofetil, rituximab, and drugs that decrease proteinuria such as angiotensin converting enzyme (ACE) inhibitors and angiotensin receptor blockers (ARBs) with inconsistent outcome. Additionally, these drugs have long-term consequences of immunosuppression and some drugs such as cyclosporine and tacrolimus affect renal function adversely when used for prolonged periods of time. (5) There is an urgent need for investigating benign therapies such as galactose. If proven to be useful, it may present a safe alternative or an adjunct to currently available therapies.

Preliminary Studies:

1. In 2008, Savin et al. showed that galactose, a simple nontoxic sugar, binds with high affinity to the FSPF in vitro.(6) They also found that trace amounts of galactose (>10-12 M) inhibited glomerular permeability activity induced by FSPF in vitro. This series of in vitro experiments also demonstrated that the effect of FSPF activity in serum can be reversed by its incubation with galactose or alternatively by pre-incubation of glomeruli with galactose. Additionally, the authors describe significantly decreased permeability activity in vivo in a single patient with post-transplant FSGS in response to both IV and oral galactose. The FSPF activity in this patient decreased progressively during the 4 weeks of galactose ingestion (from 0.8 to 0.1), and persisted 4 weeks after discontinuation of oral galactose (0.2). The proposed mechanism for this action is that FSPF have galactose-binding sites which interact with galactose of the glomerular glycocalyx, activating signal transduction in podocytes. Introduction of free galactose may block the FSPF binding sites or alter the tertiary structure of the FSPF, thus inhibiting its activity.

Despite the decrease in FSPF activity in this patient, proteinuria did not improve. The authors propose the lack of clinical response may be due to the advanced stage of kidney damage at the time of IV galactose therapy, and this patient was already on dialysis at the time of oral galactose administration.

It would be important to study the introduction of galactose early in the course of FSGS to determine if it is effective in decreasing proteinuria and delaying the progression of FSGS.

De Smet et al presented their experience with a case of 48-year old male, with nephrotic syndrome secondary to FSGS, treated with oral galactose at 10 gm BID for 6 months, at the annual meeting of American Society of Nephrology 2008 (ASN 08, TH-PO-955). Their patient had failed to respond to prednisone, cyclophosphamide, mycophenolate mofetil, cyclosporine and plasma exchanges. Prior to treatment, the FSPF was detected at 0.87 and urinary protein excretion was 4.3 gm/day. After treatment with galactose, the FSPF decreased to 0.09 and urinary protein excretion decreased to 0.56 gm/day. The success obtained in this case argues for trial in additional patients.

Methods:

1. Oral galactose therapy: After obtaining informed consent and assent FSPF will be obtained at a baseline to determine eligibility. Blood samples for FSPF will be collected in a "red-top" tube (without anti-coagulant), allowed to clot, then spin and separate. The serum will be shipped on ice for FSPF analysis to the laboratory of Virginia Savin, Medical College of Wisconsin, Milwaukee, WI. All other parameters (including weight, height, blood pressure, urinalysis, urine protein: creatinine ratio, serum albumin, creatinine, electrolytes, and glucose) will be collected at the same visit as part of standard of care. Female participants of child bearing age will be given a urine pregnancy test and excluded from the study if pregnant.

   Once patients are found to be eligible, oral galactose will be initiated at a dose of 0.2gm/kg/dose BID to a maximum of 15 gm BID for a period of 4 months. The prescribed dose of galactose powder will be dispensed to subjects in packets, mixed with 4 ounces of water, and consumed orally. FSPF will be measured again at week 16. All the other parameters will be repeated at 4, 10 and 16 weeks after starting oral galactose. Oral galactose therapy will be stopped after 16 weeks. In order to determine the clinical significance of the galactose treatment, a set of clinical parameters (weight, height, blood pressure, urinalysis, first morning urine protein: creatinine ratio, serum albumin, creatinine, electrolytes, and glucose) will be obtained at 12 weeks after discontinuation of oral galactose. Measurement of adherence with galactose will be estimated by counting the number of galactose doses returned at each subsequent monthly visit. Patients will be considered adherent if they have taken >90% of the prescribed doses.
2. Adjunct therapy of nephrotic syndrome: Each patient will remain on his or her baseline therapy immunosuppressive therapy with cyclosporine, tacrolimus or mycophenolate mofetil. Steroids dose will be tapered to 0.5mg/kg, to a maximum of 40 mg, every other day at the time of starting galactose. If patient achieves remission, as indicated by negative first morning urine for protein for 3 consecutive days, alternate day steroid therapy will be tapered by 0.12mg/kg/dose or by 10 mg/dose, once per week. If patient has sustained remission for 1 month, and is off prednisone, the dose of immunosuppressive drugs will be lowered by 25% per month until off. BP will be controlled to below 95th percentile for height. If patient is on ACE inhibitors or ARBs, the dose will stay unchanged during the duration of galactose administration unless patient is experiencing side effects of therapy. If additional therapies for control of hypertension are needed, they would be chosen from the antihypertensive drugs other than ACE inhibitors and ARBs. Diuretics will be prescribed as needed for the symptomatic relief of edema. Adjunct therapy medications described in this section are standard of care and are not for research purposes.

Result analysis:

Each patient will serve as its own control. Results will be considered clinically significant if the following criteria are met in response to oral galactose therapy at week 16 and if the reduction in urine protein: creatinine and the increase in serum albumin persist at 12 weeks after discontinuation of galactose.

1. Reduction in FSPF to <0.5 or decrease in FSPF by > 0.3
2. Decrease in first morning urine protein: creatinine ratio by 50%
3. Increase in serum albumin by >1gm/dl
4. Decrease in dose of prednisone or other immunosuppressive drugs by 25% Statistical Analysis The primary outcomes are the means of paired pre vs. post galactose treatment differences in FSPF, urine protein: creatinine ratio, serum albumin and dose of immunosuppressive drugs. We will use repeated measures ANCOVA models to estimate each primary outcome as the dependent variable while holding constant pre-treatment levels. Therefore, the independent variable will be the pre-treatment level of the corresponding dependent variable, The model will be used to estimate the mean difference +/- the 95% confidence interval (CI) corresponding to the mean level of the dependent variable at pre-treatment. We will consider the pre-post difference to be statistically significant if the 95% CI around the result fails to include 0 and to be clinically significant if it meets the criteria specified above.

Adequacy of the Sample: We evaluated the effect size difference that could be detected with 80% and 90% power in a pre-post treatment study of galactose involving 10 patients assessed pre-treatment and post-treatment. The correlation between measurements on the same person was assumed to be .7 and the two-tailed type 1 error was set at 0.05. The study will have better than 90% power to detect effect size differences of 0.6 sd and better than 80% power to detect effect size differences of 0.5 sd. These are considered to be moderate effect sizes.

Research Facilities: The FS permeability factor will be tested in the laboratory of Virginia Savin MD (Center for Glomerular Pathophysiology, Medical College of Wisconsin, Milwaukee, WI) using previously described methods.(7)

Risks and Side Effects:

FSGS is a difficult to treat disease associated with poor outcomes, including progression to end stage renal disease. Galactose is a naturally occurring simple sugar and oral galactose supplementation has no known side risks or side effects in humans. Patients eligible for this study are those who have failed to respond to the current alternative treatments for FSGS, which include steroids and other immunosuppressive agents, such as cyclosporine, tacrolimus, mycophenolate mofetil, and rituximab. These alternative immunosuppressive treatments have many long term complications, some of which include stunted growth, nephrotoxicity, hyperlipidemia, and diabetes. There is an urgent need for investigating benign therapies such as galactose, which may present a safe alternative or an adjunct to current therapies.

There are no known side effects of oral galactose supplementation and no reports of toxicity with chronic use in humans. The Certificate of Origin for the D-Galactose product from FerroPfanstiehl is included in the Appendix and certifies that the D-Galactose to be used in our study is safe for human consumption.

D-Galactose is administered safely in diagnostic testing for both glycogen storage disease and cirrhotic liver disease (8) and as sonographic contrast agents, such as Levovist ® (Bayer). Galactose has also been successfully administered as a treatment in Fabry's disease. (9) In this case report, IV galactose infusions were administered at a dose of 1 g/kg every other day for 2 years during which time liver function tests remained normal. Possible associations between dairy intake and ovarian cancer has been investigated with inconclusive results. A 2006 pooled analysis of 12 cohort studies done by Harvard School of public health found no association of intake of dairy foods with ovarian cancer and a statistically insignificant increase in risk of ovarian cancer at intakes of lactose > 30 g/d. This study involved analyzing surveys of reported dairy intake, but did not account for the presence of other factors in milk, such as hormones, that could contribute to ovarian cancer risk (10). Another 2005 meta-analysis in the European Journal of Cancer Prevention found no association between milk/dairy products or galactose metabolism and ovarian cancer risk. (11) In addition to occurring naturally in milk, galactose has been approved by the FDA as a substance Generally Recognized as Safe (GRAS) as an ingredient in infant formula and other baby foods and pediatric nutrition supplements in the form of galacto-oligosaccharides (a compound made of 1 to 7 galactose molecules linked to a glucose molecule at the reducing end). (www.fda.gov/food/foodingredientspackaging/generallyrecognizedassafeGRAS/GRASListings/ucm153910.htm)

Benefits:

FSGS is resistant to steroid therapy and many other immunosuppressive drugs, and is associated with poor outcome. Approximately 50% of patients with FSGS progress to ESRD within 5-10 years and in about 30% of children, FSGS can recur after transplantation.(1) Given the devastating course of this disease and the benign nature of the proposed galactose treatment, the anticipated benefits far outweigh the risks. If effective, galactose supplementation could stop the progression of FSGS, limiting glomerular damage and preventing progression of the disease to ESRD. The potential benefit of preserving kidney function and preventing the need for dialysis or transplantation is significant for both participants in this study and for other children with FSGS who may benefit from galactose therapy in the future.

ELIGIBILITY:
Inclusion Criteria:

1. 2-21 years old
2. Biopsy proven FSGS or minimal change with steroid resistance
3. Presence of FSPF (defined as permeability activity >0.5)
4. Presence of nephrotic range proteinuria (urine protein: creatinine ratio >2) at the time of enrollment.
5. Persistent nephrotic range proteinuria despite being on stable immunosuppressive medications (cyclosporine, tacrolimus or mycophenolate mofetil) for at least 12 weeks and/or persistent nephrotic range proteinuria despite being on stable dose of angiotensin converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARBs) for 12 weeks.
6. Stable serum creatinine (change of less than 0.3 mg/dl) in the prior 3 months.
7. Schwartz estimated (e) glomerular filtration rate (GFR) >60ml/min/1.73m2

Exclusion Criteria:

1. Secondary FSGS
2. Onset of nephrotic syndrome in infancy.
3. Presence of acute renal failure (as defined by acute kidney injury criteria) at the time of enrollment. These children can be enrolled 1 month after resolution of acute renal failure (ARF).
4. Decreasing renal function (persistent increase in serum creatinine of greater than 0.3 mg/dl over baseline in the prior 3 months).
5. Use of another investigational drug
6. Pregnant or unable to comply with contraceptive measures in females of child bearing age
7. eGFR < 60 ml/min per 1.73 m2
8. Children with Galactosemia
9. Children with type 1 or 2 diabetes

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2009-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asha Moudgil, MD, Principal Investigator — Children's National Research Institute; Kristen Sgambat, MS, RD, Study Director — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Fine RN. Recurrence of nephrotic syndrome/focal segmental glomerulosclerosis following renal transplantation in children. Pediatr Nephrol. 2007 Apr;22(4):496-502. doi: 10.1007/s00467-006-0361-6. Epub 2006 Dec 21. PMID 17186280
- [Background] Srivastava T, Simon SD, Alon US. High incidence of focal segmental glomerulosclerosis in nephrotic syndrome of childhood. Pediatr Nephrol. 1999 Jan;13(1):13-8. doi: 10.1007/s004670050555. PMID 10100283
- [Background] Tryggvason K, Patrakka J, Wartiovaara J. Hereditary proteinuria syndromes and mechanisms of proteinuria. N Engl J Med. 2006 Mar 30;354(13):1387-401. doi: 10.1056/NEJMra052131. No abstract available. PMID 16571882
- [Background] Trachtman H, Greenbaum LA, McCarthy ET, Sharma M, Gauthier BG, Frank R, Warady B, Savin VJ. Glomerular permeability activity: prevalence and prognostic value in pediatric patients with idiopathic nephrotic syndrome. Am J Kidney Dis. 2004 Oct;44(4):604-10. PMID 15384010
- [Background] Burdmann EA, Andoh TF, Yu L, Bennett WM. Cyclosporine nephrotoxicity. Semin Nephrol. 2003 Sep;23(5):465-76. doi: 10.1016/s0270-9295(03)00090-1. PMID 13680536
- [Background] Savin VJ, McCarthy ET, Sharma R, Charba D, Sharma M. Galactose binds to focal segmental glomerulosclerosis permeability factor and inhibits its activity. Transl Res. 2008 Jun;151(6):288-92. doi: 10.1016/j.trsl.2008.04.001. Epub 2008 May 2. PMID 18514139
- [Background] Savin VJ, Sharma R, Sharma M, McCarthy ET, Swan SK, Ellis E, Lovell H, Warady B, Gunwar S, Chonko AM, Artero M, Vincenti F. Circulating factor associated with increased glomerular permeability to albumin in recurrent focal segmental glomerulosclerosis. N Engl J Med. 1996 Apr 4;334(14):878-83. doi: 10.1056/NEJM199604043341402. PMID 8596570
- [Background] Shreeve WW, Shoop JD, Ott DG, McInteer BB. Test for alcoholic cirrhosis by conversion of [14C]- or [13C]galactose to expired CO2. Gastroenterology. 1976 Jul;71(1):98-101. PMID 1278655
- [Background] Frustaci A, Chimenti C, Ricci R, Natale L, Russo MA, Pieroni M, Eng CM, Desnick RJ. Improvement in cardiac function in the cardiac variant of Fabry's disease with galactose-infusion therapy. N Engl J Med. 2001 Jul 5;345(1):25-32. doi: 10.1056/NEJM200107053450104. No abstract available. PMID 11439944
- [Background] Genkinger JM, Hunter DJ, Spiegelman D, Anderson KE, Beeson WL, Buring JE, Colditz GA, Fraser GE, Freudenheim JL, Goldbohm RA, Hankinson SE, Koenig KL, Larsson SC, Leitzmann M, McCullough ML, Miller AB, Rodriguez C, Rohan TE, Ross JA, Schatzkin A, Schouten LJ, Smit E, Willett WC, Wolk A, Zeleniuch-Jacquotte A, Zhang SM, Smith-Warner SA. A pooled analysis of 12 cohort studies of dietary fat, cholesterol and egg intake and ovarian cancer. Cancer Causes Control. 2006 Apr;17(3):273-85. doi: 10.1007/s10552-005-0455-7. PMID 16489535
- [Background] Qin LQ, Xu JY, Wang PY, Hashi A, Hoshi K, Sato A. Milk/dairy products consumption, galactose metabolism and ovarian cancer: meta-analysis of epidemiological studies. Eur J Cancer Prev. 2005 Feb;14(1):13-9. doi: 10.1097/00008469-200502000-00003. PMID 15677891
- [Background] Schwartz GJ, Haycock GB, Edelmann CM Jr, Spitzer A. A simple estimate of glomerular filtration rate in children derived from body length and plasma creatinine. Pediatrics. 1976 Aug;58(2):259-63. PMID 951142
- [Background] De Smet E, Rioux JP, Ammann H, Deziel C, Querin S. FSGS permeability factor-associated nephrotic syndrome: remission after oral galactose therapy. Nephrol Dial Transplant. 2009 Sep;24(9):2938-40. doi: 10.1093/ndt/gfp278. Epub 2009 Jun 9. PMID 19509024

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Galactose
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Galactose
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.7 (4)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Focal Segmental Glomerulosclerosis Permeability Factor (FSPF)
Description: FSPF is reported in relation to its induction of glomerular albumin permeability (Palb) of isolated glomeruli on a range from 0 to 1, with 0 indicative of normal glomeruli and 1 indicative of injury to the permeability barrier. Results will be considered clinically significant if the following criteria is met in response to oral galactose therapy at week 16: Reduction in FSPF to <0.5 Palb or decrease in FSPF by > 0.3 Palb.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Palb
Arm/Group | Galactose
Number analyzed (Participants) | 7
Palb
  Baseline FSPF | 0.69 (0.11)
  16 Week FSPF | 0.35 (0.21)
Statistical Analysis 1: Comparison: Galactose; Test type: Superiority or Other; p = 0.009, t-test, 2 sided — p value reflects the difference in mean FSPF pre vs post galactose treatment

2. Secondary Outcome: Number of Participants Achieving Complete or Partial Remission at 16 Weeks
Description: Results will be considered clinically significant if the following criteria is met in response to oral galactose therapy at week 16. Complete remission is defined as (Urine Protein:Creatinine ratio [UPC] <0.2 g/g). Partial remission is defined as UPC 0.2-2 g/g.
Time Frame: 16 weeks
Measure: Number; unit: participants in remission at 16 weeks
Arm/Group | Galactose
Number analyzed (Participants) | 7
participants in remission at 16 weeks | 0

ADVERSE EVENTS:
Time Frame: Monthly for duration of galactose therapy (4 months)
Arm/Group | Galactose
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galactose (N=7)
Diarrhea (Gastrointestinal disorders) | 1 (1) — 1 subject experienced diarrhea, but also taking other medications known to have side effect of diarrhea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes